CLINICAL TRIAL: NCT02352532
Title: Using Structural Health Monitoring to Improve Diagnosis and Treatment of Low Back Injury in U.S. Service Members- Phase 2
Acronym: SWE/DN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Collaborators: Telemedicine & Advanced Technology Research Center (TATRC) (Unknown); Army Medical Department Center and Schools (Unknown)
Responsible Party: Principal Investigator, Shane Koppenhaver, PT, PhD, Baylor University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: #10586012
Record Dates: First submitted 2015-01-26; First posted 2015-02-02 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Low Back Pain
Keywords: Dry Needling; Shear Wave Elastography; Ultrasound
MeSH Terms: conditions — Low Back Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Back Pain - Dry Needling (Experimental)
  Interventions: Other: Dry Needling
- Low Back Pain - Sham (Sham Comparator)
  Interventions: Other: Sham Needling
- Asymmptomatic - Dry Needling (Active Comparator)
  Interventions: Other: Dry Needling

INTERVENTIONS:
Other: Dry Needling — The dry-needling treatment will consist of inserting a sterile needle into needling the prone participant's lumbar multifidus and paraspinal muscles, 1-2 times each, in regions of local tenderness to palpation and/or regions with palpable trigger points. All needling treatment will be performed with FDA approved (FDA regulation # 880.5580) disposable 0.30 x 50-60 mm stainless steel Seirin J-type needles (Seirin, Japan). Each needle insertion will last approximately 5 seconds using a "pistoning" (in and out) technique.
  Other Names: Trigger point dry needling
  Arms: Asymmptomatic - Dry Needling; Low Back Pain - Dry Needling
Other: Sham Needling — The sham dry-needling procedure will mimic the dry needling procedures by placing a sharp object in a needling guide tube against the skin (see figure). The sharp object will be rocked and twisted to simulate treatment, but will not pierce the skin. We have used this sham dry-needling technique in a previous study performed at AMEDDC&S and have found it to be indistinguishable from real dry needling by the great majority of participants.
  Arms: Low Back Pain - Sham

SUMMARY:
The focus of this project is to evaluate the diagnostic utility of Shear Wave Elastography (SWE) in individuals after routine low back injury and begin an initial investigation of it's ability to effectively guide physical therapy treatment with dry-needling as a relevant treatment intervention.

Specific Aim #1: Evaluate the diagnostic utility of SWE in differentiating individuals with and without LBP. The investigators will also examine the interaction between tissue change and clinical improvement. The investigators hypothesize that individuals with LBP will have higher muscle stiffness (shear modulus) at rest and impaired (lower) stiffness during contraction than individuals without LBP.

Specific Aim #2: Evaluate the effectiveness of dry-needling in decreasing aberrant muscle stiffness in individuals with LBP. The investigators hypothesize that individuals with LBP that receive dry-needling will exhibit larger changes than both individuals with LBP that receive sham dry-needling and than individuals without LBP that receive dry-needling.

Specific Aim #3: Evaluate the effectiveness of dry-needling in decreasing pain and disability in individuals with LBP. The investigators hypothesize that individuals with LBP that receive dry-needling will exhibit larger improvements than individuals with LBP that receive sham dry-needling.

DETAILED DESCRIPTION:
Low back pain (LBP) is the second most frequent reason for health care visits and a leading cause of medical evacuation from theater. Traditional medical diagnosis based on static imaging strategies (e.g. MRI) has failed to improve management of this epidemic. Functional assessment of lumbar musculature using ultrasound imaging provides evidence of clinically relevant deficits in the lumbar multifidus (LM) muscle of patients with LBP, however such procedures are likely only valid within a narrow range of assessment conditions. Shear-Wave Elastography (SWE) is an evolving non-invasive ultrasound imaging technology capable of quantifying tissue stiffness (i.e., elasticity). Originally developed to improve diagnosis of soft tissue tumors, SWE is beginning to be used to as an alternative and more stable method of functional assessment of muscles.

This study will be the second project in a line of research aimed at improving the diagnosis, management, and treatment of patients with LBP using a new structural health monitoring technique called shear wave elastography (SWE). Since no previous studies had used SWE in the lumbar multifidus muscle, the initial project developed the measurement technique to be used with this device. We also established normative parameters, variance, and reliability estimates of SWE outcomes in asymptomatic individuals. A previous study, also performed at AMEDDC&S, found that individuals with LBP whom received dry needling to the lumbar multifidus muscle exhibited a reduction in pain and disability that was associated with an improved ability to contract the lumbar multifidus. The focus of this second project is to evaluate the diagnostic utility of SWE in individuals after routine low back injury and begin an initial investigation of it's ability to effectively guide physical therapy treatment with dry-needling as a relevant treatment intervention.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 18 - 65 years
* Read and speak English well enough to provide informed consent and follow study instructions
* Active duty military or DOD beneficiary
* History of prior surgery to the lumbosacral spine
* Received manual therapy, acupuncture, or dry-needling interventions to the lumbosacral spine within the past 4 weeks
* Currently taking anticoagulant medications or those individuals with a medical history of bleeding disorder
* History of systemic inflammatory disease or other serious spinal pathology (e.g. annular tears of the intervertebral disc, spinal stenosis, fracture)
* Known pregnancy and/or inability to lie prone and fully elevate bilateral arms
* Presence of neurogenic LBP defined by either a positive ipsilateral or contralateral straight leg raise (reproduction of symptoms at <45°) or reflex, sensation, or strength deficits in a pattern consistent with nerve root compression
* Medical "red flags" of a potentially serious condition including cauda equina syndrome, major or rapidly progressing neurological deficit, fracture, cancer, infection, or systemic disease

Exclusion Criteria:

* History of prior surgery to the lumbosacral spine
* Received manual therapy, acupuncture, or dry-needling interventions to the lumbosacral spine within the past 4 weeks
* Currently taking anticoagulant medications or those individuals with a medical history of bleeding disorder
* History of systemic inflammatory disease or other serious spinal pathology (e.g. annular tears of the intervertebral disc, spinal stenosis, fracture)
* Known pregnancy and/or inability to lie prone and fully elevate bilateral arms
* Presence of neurogenic LBP defined by either a positive ipsilateral or contralateral straight leg raise (reproduction of symptoms at <45°) or reflex, sensation, or strength deficits in a pattern consistent with nerve root compression
* Medical "red flags" of a potentially serious condition including cauda equina syndrome, major or rapidly progressing neurological deficit, fracture, cancer, infection, or systemic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in muscle stiffness and activation utilizing shear-wave elastography after dry needling - one week follow-up | 7 days
  SWE images of the lumbar multifidus and paraspinal muscles will be acquired at rest and during sub-maximal isometric contraction. All SWE images will be obtained using a Supersonic Aixplorer ultrasound system with a 50mm 10-2 MHz linear array. The sub-maximal contraction of the lumbar multifidus will be elicited by a contralateral arm lift maneuver while holding a small hand weight following techniques outlined in our previous work.42 The weight used will depend on the participant's body weight and will elicit approximately 30% of the MVC of the lumbar multifidus muscle as previously shown by fine wire EMG.43 Participants weighing less than 68 kg (150 lbs) will use .68 kg (1.5 lbs), those between 68-90 kg (150-200 lbs) will use .91 kg (2 lbs), and those greater than 91 kg (200 lbs) will use 1.36 kg (3 lbs). Participants will be instructed as follows: "lift your arm approximately 2 inches (5 cm) off the table".
Change in pain pressure threshold utilizing pressure algometry after dry needling | 5 minutes
  Pressure algometry will used in the current study to determine the most painful spinal level at baseline and as a secondary outcome measure, pain pressure threshold (PPT), to assess abnormalities in nociceptive processing or hyperalgisia 37,38. PPT measures have been found to be highly reliable,39-41 especially when taken by the same rater (ICC=0.94-.097) 40. A digital pressure algometer (Wagner Force Ten FDX, Wagner Instruments, Greenwich, CT) will be used to measure PPT in the lumbar multifidus and paraspinal muscles on the side that the participant reported as more symptomatic. The pressure algometer will held by the examiner directly perpendicular to the muscle belly, approximately 1.5 cm lateral to the spinous process. The algometer will be advanced at a rate of approximately 5N/sec. and participants are instructed to verbally signal when they first perceive the force exerted as painful. PPT at each location will taken three times and averaged to reduce variability.
  Pressure
Change in muscle stiffness and activation utilizing shear-wave elastography after dry needling. | 5 minutes
  SWE images of the lumbar multifidus and paraspinal muscles will be acquired at rest and during sub-maximal isometric contraction. All SWE images will be obtained using a Supersonic Aixplorer ultrasound system with a 50mm 10-2 MHz linear array. The sub-maximal contraction of the lumbar multifidus will be elicited by a contralateral arm lift maneuver while holding a small hand weight following techniques outlined in our previous work.42 The weight used will depend on the participant's body weight and will elicit approximately 30% of the MVC of the lumbar multifidus muscle as previously shown by fine wire EMG.43 Participants weighing less than 68 kg (150 lbs) will use .68 kg (1.5 lbs), those between 68-90 kg (150-200 lbs) will use .91 kg (2 lbs), and those greater than 91 kg (200 lbs) will use 1.36 kg (3 lbs). Participants will be instructed as follows: "lift your arm approximately 2 inches (5 cm) off the table".
Change in pain pressure threshold utilizing pressure algometry after dry needling - 1 week follow-up | 7 days
  SWE images of the lumbar multifidus and paraspinal muscles will be acquired at rest and during sub-maximal isometric contraction. All SWE images will be obtained using a Supersonic Aixplorer ultrasound system with a 50mm 10-2 MHz linear array. The sub-maximal contraction of the lumbar multifidus will be elicited by a contralateral arm lift maneuver while holding a small hand weight following techniques outlined in our previous work.42 The weight used will depend on the participant's body weight and will elicit approximately 30% of the MVC of the lumbar multifidus muscle as previously shown by fine wire EMG.43 Participants weighing less than 68 kg (150 lbs) will use .68 kg (1.5 lbs), those between 68-90 kg (150-200 lbs) will use .91 kg (2 lbs), and those greater than 91 kg (200 lbs) will use 1.36 kg (3 lbs). Participants will be instructed as follows: "lift your arm approximately 2 inches (5 cm) off the table".

SECONDARY OUTCOMES:
Change in Numerical Pain Rating Scale | 7 days
  The numeric pain rating scale (NPRS) will be used to assess the participant's pain levels. The participant will grade his/her pain on an 11-point scale ranging from 0 (no pain) to 10 (worst imaginable pain).The NPRS has been shown to be a reliable, generalizable, and internally consistent measure of clinical and experimental pain intensity in individuals with musculoskeletal disorders.33,34 A 2-point change on the NPRS is required to be clinically meaningful.
Change in function and disability utilizing a physical exam | 7 days
  Participants with current LBP will undergo a standardized clinical examination based the Treatment Based Classification System.31 Patients without current LBP will undergo an abbreviated examination primarily focused on sociodemographic
Change in Oswestry Disability Index | 7 days
  The Oswestry Disability Index (ODI) is a LBP-specific subjective measure of disability. Users are asked to rate the difficulty of performing 10 functional tasks on a scale of 0 to 5 with different descriptors for each task. A total score out of 100 is calculated by summing each score and doubling the total. The answers provide a score between 0 and 100, with higher scores representing more disability. It has been shown to have excellent test-retest reliability (ICC2,1=.90), good validity, and superior responsiveness compared to other leading disability scales.32

OTHER OUTCOMES:
Global Rate of Change | 7 days
  The global rating of change (GRC) assesses subjective perception of overall change and the importance of that change. A 15-point Likert type scale ranging from -7 (very great deal worse) to +7 (a very great deal better) and a 6-point Likert type scale ranging from 1 (a tiny bit important) to 6 (a very great important) will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Army Medical Department Center and Schools, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided